CLINICAL TRIAL: NCT00154232
Title: A 3 Month, Multicenter, Open-label Study to Evaluate the Impact of the Immunosuppressive Combination of Enteric-Coated Mycophenolate Sodium (EC- MPS), Basiliximab and Cyclosporine for Microemulsion With C2 Monitoring, on Efficacy and Safety Outcomes in de Novo Kidney Transplant Recipients at Potential High Risk of DGF.
Brief Title: Study to Evaluate the Combination of Enteric-coated Mycophenolate Sodium (EC-MPS), Basiliximab, and C2-monitored Cyclosporine in de Novo Renal Transplant Recipients at Potential High Risk of Delayed Graft Function (DGF)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CERL080AAR01
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-11

CONDITIONS: Renal Transplantation
Keywords: Renal transplantation, DGF, basiliximab, EC-MPS, cyclosporine

INTERVENTIONS:
Drug: Enteric-Coated Mycophenolate Sodium (EC-MPS)

SUMMARY:
The aim of the study is to assess the short-term benefit of the combination of basiliximab, EC-MPS and cyclosporine microemulsion with C2 monitoring on the prophylaxis of acute rejection in a population of de novo renal transplant patients at potential high risk of DGF.

ELIGIBILITY:
Inclusion Criteria:

- Age 18-70 years old

* Patients receiving a primary or secondary cadaveric or living donor kidney
* Patients who have given written informed consent for study participation
* Females capable of becoming pregnant must have a negative pregnancy test at baseline and are required to practice birth control for the duration of the study and at least for four months following the last dose of basiliximab.

Exclusion Criteria:

* Recipient of multi-organ transplants or previously transplanted organs other than kidney
* Recipient of dual kidney transplants
* Recipient of a transplanted kidney from a Non-Heart Beating Donor (NHBD)
* Recipient of a HLA identical living-donor kidney
* Patients with a PRA level (past or current level) greater than 20%
* Patients anticipated by investigators to require induction therapy with OKT3, ATGAM, or Thymoglobulin for any reason
* Patients with any medical condition which, in the opinion of the investigator, would preclude the patient from participating in the study
* Cold ischemia time larger than 36 hours.
* Patients who have received an investigational drug or therapy within one month prior to study entry or if such therapy is to be instituted post-transplantation.
* Female transplant candidates who are pregnant, lactating, or of childbearing potential and not willing to practice an acceptable method of contraception
* Patients with a known hypersensitivity to cyclosporine
* Patients with a known malignancy or a history of malignancy, other than successfully treated non-metastatic basal or squamous cell carcinoma of the skin
* Known HIV positive antibody status
* Evidence of any clinically relevant (per investigator determination) active infection
* Patients unable to participate in the study for the full 3-month study period
* Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 46
Dates: Start 2004-06; Primary Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Incidence of first episodes of BPAR at month 3 post transplant

SECONDARY OUTCOMES:
Incidence of patients death at month 3 post transplant.
Incidence of graft loss or, synonymously, graft failure)
The allograft will defined as lost (or: to have failed)
when the patient begins dialysis treatments without
subsequent graft recovery.
The time of graft failure will be defined as the time of start of dialysis, or time of nephrectomy, whatever occurs first.
Number of myfortic dose adjustments/discontinuations

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis